CLINICAL TRIAL: NCT01136954
Title: An Open-label Extension Study Following a Double-blind, Randomized, Placebo-controlled, Multi-centre Study to Assess the Efficacy and Safety of Adjunctive Zonisamide in Pediatric Partial Onset Seizures
Brief Title: A Study to Assess the Efficacy and Safety of Adjunctive Zonisamide in Paediatric Partial Onset Seizures (CATZ Extension Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2090-E044-313; 2007-000198-53 (EudraCT Number)
Record Dates: First submitted 2010-05-26; First posted 2010-06-04 (Estimated); Results first posted 2013-02-06 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2015-11

CONDITIONS: Partial Seizures
MeSH Terms: conditions — Seizures | interventions — Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Zonisamide

INTERVENTIONS:
Drug: Zonisamide — Transition Period from Study E2090-E044-312: Placebo Open-Label Period: 1 to 8 mg/kg orally per day for approximately 59 weeks.
  Other Names: Zonegran

SUMMARY:
The purpose of this study is to assess the long-term safety and efficacy of zonisamide used as an adjunctive treatment in pediatric subjects treated with 1 or 2 other anti-epileptic drugs (AEDs).

DETAILED DESCRIPTION:
Those subjects who completed the double-blind study (E2090-E044-312) will be invited to participate in this extension study. The study consists of two main parts: Transition Period (double-blind) and Open Label Period. The study will start with the Transition Period during which subjects already on zonisamide will continue on the same dose of zonisamide and those who were taking placebo will be up-titrated to an appropriate dose of zonisamide. After all subjects have completed the Transition Period, the study will become open-label with every subject on the study receiving zonisamide. The study medication will be taken once daily in the evening. For those subjects previously in the placebo group, dosing with zonisamide will start with a dose of approximately 1 mg/kg. In order that the blind is maintained from the previous study, these subjects will initially continue taking the same number of placebo capsules as they were taking in the Maintenance Period of the E2090-E044-312 study until the up- titration is completed. Those subjects previously in the zonisamide arm will continue on the same dose which they received during the Maintenance Period of the E2090-E044-312 study. In order that the blind is maintained, they will also take placebo capsules in order to mirror the up- titration dose regimen of the subjects previously randomized to receive placebo in the E2090-E044-312 study. All subjects will stop taking placebo capsules after the Transition Period is complete. The duration of the Transition Period depends on the dose the subject appeared to have received when completing the core study E2090-E044-312. For those who completed on 8 mg/kg, the Transition Period will last 7 weeks. For those on 6 mg/kg, the Transition Period will last 5 weeks. However, during the double-blind Transition Period, some subjects may experience adverse events (AEs). If this should occur, the subject may be down titrated to one level above the minimal dose. The overall duration of the study will be up to 59 weeks. The overall duration of the Transition Period may thus be as short as 2 weeks or prolonged to as many as 11 weeks.

The Open Label Period will continue for up to a maximum of 59 weeks (approximately 15 months).

At the end of the study, Eisai will continue to supply zonisamide as part of this open-label extension protocol until the marketing authorisation of zonisamide for this indication or further development in this indication is stopped. In countries where no marketing authorisation will be applied for, Eisai has a compassionate use policy which can be applied for, if required.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Subject has completed the double-blind study E2090-E044-312.
2. Parent/caregiver is willing to sign an informed consent where the subject is under the age of consent.
3. Subject is male or female aged 6 to 18 years who is willing to give informed (written or verbal) assent, if applicable. If mandated by local regulations, subjects of relevant age will be required to sign an appropriate informed consent.
4. Subject is in general good health as determined by medical history, physical exam and screening laboratory results.

EXCLUSION CRITERIA:

1. Subject has a body weight < 20 kg.
2. Subject has developed a history of renal calculi or renal insufficiency (creatinine level > 135 µmol/l (1.5 mg/dl).
3. Subject has a known diagnosis of human immunodeficiency virus (HIV) or hepatitis B or C.
4. Subject has a history of sensitivity to sulfonamide drugs or zonisamide and its excipients.
5. Female subject of 10 years of age or greater, or of child bearing potential (i.e. started menses) and is not taking or prepared to take a medically acceptable form of contraception (i.e. oral contraceptive pill, surgical sterilization, an implant or injected form of contraception, or intrauterine device), or who is not prepared to abstain from sexual activity for the duration of the study and for one month after the last administration of study medication. NOTE: Should a female subject become of child bearing potential during the study, they must be reconsented in order to given consent to undergo pregnancy testing and either confirm abstinence or receive a medically appropriate form of contraception.
6. Subject has a recent history of excessive alcohol use or drug abuse.
7. Subject has a history of suicide attempt.
8. Subject has a clinically significant organic disease.
9. Subject has a history of demonstrated non-compliance with treatment or subject or parent/legal guardian can be reasonably expected not to be compliant with study procedures or to complete the study.
10. Frequent need of rescue benzodiazepines (one or more times a month).
11. Concomitant use of acetazolamide, carbonic anhydrase inhibitors such as topiramate, furosemide and drugs with anticholinergic activity.
12. Concomitant use of felbamate or use of felbamate within 2 months prior to Visit 1 of the E2090-E044-312 study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2008-07; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rob van Maanen, M.D., MFPM, Study Director — Eisai Limited
Locations (1):
- Firenze, 50132, FI, Italy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who completed E2090-E044-312 (NCT00566254)"Study 312" core study were invited to participate in this extension study.
Groups:
- Zonisamide(Placebo During Core Study): Participants previously receiving placebo in Study 312, started dosing with zonisamide with a dose of 1 mg/kg/day and titrated upwards with weekly dose increases until a dose of 8 mg/kg/day was reached at the end of the Transition Period (weeks 2 -11). Downtitration was allowed between the limits of 1 to 8 mg/kg/day during Transition Period. Subsequently, a 45-57 week Open-label period followed. Placebo dosing ceased in Open-label Period.
- Zonisamide (Zonisamide During Core Study): Participants previously receiving zonisamide in Study 312 continued taking the same dose of study drug (8 mg/kg/day),supplemented with an increasing number of placebo capsules to mirror the up-titration regimen being followed by those previously receiving placebo.Down-titration was allowed between the limits of 1 to 8 mg/kg/day during Transition Period.Subsequently, a 45-57 week Open-label period followed.
Period: Overall Study
Arm/Group | Zonisamide(Placebo During Core Study) | Zonisamide (Zonisamide During Core Study)
Started | 72 | 72
Completed | 48 | 51
Not Completed | 24 | 21
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lack of Efficacy | 14 | 13
Not completed — Physician Decision | 0 | 1
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide(Placebo During Core Study) | Zonisamide (Zonisamide During Core Study) | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Customized [Number; unit: Participants]
  6-11 Years | 34 | 33 | 67
  12-18 Years | 38 | 39 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 41 | 73
  Male | 40 | 31 | 71

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Non-Serious Adverse Events With Greater Than 5% Frequency
Description: Treatment Emergent Adverse Event (TEAE) is defined as an Adverse Event with a start date on or after Day 1 and within 15 days of last dose. For each event, each participant experiencing an event is only counted once even if they had multiple episodes.
Time Frame: Week 1 through Week 59
Population: Safety Population (all subjects who entered the study and received at least one dose of study drug)
Measure: Number; unit: Participants
Groups:
- Zonisamide (Placebo During Core Study): Participants previously receiving placebo in Study 312, started dosing with zonisamide with a dose of 1 mg/kg/day and titrated upwards with weekly dose increases until a dose of 8 mg/kg/day was reached at the end of the Transition Period (weeks 2 -11). Downtitration was allowed between the limits of 1 to 8 mg/kg/day during Transition Period. Subsequently, a 45-57 week Open-label period followed. Placebo dosing ceased in Open-label Period.
Arm/Group | Zonisamide (Placebo During Core Study) | Zonisamide (Zonisamide During Core Study)
Number analyzed (Participants) | 72 | 72
Participants
  Nasopharyngitis | 6 | 9
  Bronchitis | 4 | 3
  Respiratory tract infection | 2 | 4
  Headache | 4 | 7
  Weight decreased | 6 | 6
  Abdominal pain | 1 | 4
  Decreased Appetite | 5 | 4

2. Secondary Outcome: Percentage of Participants With a Decrease From Baseline in 28-day Seizure Frequency of =50%(Responder) in the Open Label Period
Description: A participant with a decrease from baseline in seizure frequency of =50 % was considered a responder. Participants'parent or guardian maintained a seizure diary recording the date,number, and type of seizures the subject had. The primary analysis assessed the percent of responders from baseline in the Open Label Visit Period. Seizure frequency of simple partial, complex partial, and partial seizures with secondary generalization were assessed.
Time Frame: Baseline through Week 59
Population: Safety Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Zonisamide(Placebo During Core Study) | Zonisamide (Zonisamide During Core Study)
Number analyzed (Participants) | 72 | 72
Percentage of Participants | 55.6 | 56.9

3. Secondary Outcome: Median Change From Study 312 Baseline in the 28-day Seizure Frequency During the Open Label Period
Description: Participants' parent or guardian maintained a seizure diary recording the date, number, and type of seizures the subject had. Seizure frequency of simple partial, complex partial, and partial seizures with secondary generalization were assessed from baseline of study 312 through the Open Label Visit Period.
Time Frame: Baseline of study 312 (Week -8 to Week 0) to Week 59 of study 313
Population: Safety Population
Measure: Median (Full Range); unit: Seizures
Arm/Group | Zonisamide(Placebo During Core Study) | Zonisamide (Zonisamide During Core Study)
Number analyzed (Participants) | 72 | 72
Seizures | -3.8 [-89 to 73] | -4.7 [-95 to 50]

4. Secondary Outcome: Median Percent Change From Study 312 Baseline in the 28-day Seizure Frequency During the Open Label Period
Description: Participants' parent or guardian maintained a seizure diary recording the date, number, and type of seizures the subject had. Seizure frequency of simple partial, complex partial, and partial seizures with secondary generalization were assessed from baseline of study 312 through the Open Label Visit Period. Percentage change = 100% x (seizure frequency at period - seizure frequency at Study 312 baseline)/seizure frequency at Study 312 baseline.
Time Frame: Baseline of study 312 (Week -8 to Week 0) to Week 59 of study 313
Population: Safety Population
Measure: Median (Full Range); unit: Percentage Change
Arm/Group | Zonisamide(Placebo During Core Study) | Zonisamide (Zonisamide During Core Study)
Number analyzed (Participants) | 72 | 72
Percentage Change | -64.6 [-100 to 174] | -67.9 [-100 to 262]

ADVERSE EVENTS:
Time Frame: "Treatment-Emergent Adverse Events (TEAE) were collected, and includes all Adverse Events (AE) with a start date on or after Day 1 and within 15 Days of last dose, including AEs with missing start dates. Participants were followed for up to 61 weeks.
Description: Treatment-emergent AEs were summarized by period (Transition, Open-label, Down-titration), treatment group,body system, and preferred term (PT).
Arm/Group | Zonisamide(Placebo During Core Study) | Zonisamide (Zonisamide During Core Study)
Serious Adverse Events (participants affected / at risk) | 3/72 | 7/72
Other Adverse Events (participants affected / at risk) | 18/72 | 25/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide(Placebo During Core Study) (N=72) | Zonisamide (Zonisamide During Core Study) (N=72)
Bronchitis (Infections and infestations) | 0 | 1
Lymph gland infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 0 | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Foreign body aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide(Placebo During Core Study) (N=72) | Zonisamide (Zonisamide During Core Study) (N=72)
Nasopharyngitis (Infections and infestations) | 6 | 9
Bronchitis (Infections and infestations) | 4 | 3
Respiratory tract infection (Infections and infestations) | 2 | 4
Headache (Nervous system disorders) | 4 | 7
Weight decreased (Investigations) | 6 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 4
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No